CLINICAL TRIAL: NCT05352139
Title: Prospective Multi-Center Patient Registry for Patients With Elbow, Hip, and Calcific Shoulder Tendinosis Treated Utilizing the TenJet Hydroresection System
Brief Title: Treatment of Tendinosis Using the TenJet Hydroresection System
Status: Enrolling by invitation | Type: Observational
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: WIRB CMEH 01
Record Dates: First submitted 2022-04-25; First posted 2022-04-28 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Tendinopathy; Tendinosis
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Elbow Tendinosis (Epicondylitis): Treatment of participants who present with either lateral or medial epicondylitis
  Interventions: Procedure: Resection (removal) of the degenerative tissue using the Hydrocision TenJet system; Device: Hydrocision Tenjet System
- Hip Tendinosis (Gluteal Tendinopathy): Treatment of participants diagnosed with Recalcitrant Gluteal Tendinopathy
  Interventions: Procedure: Resection (removal) of the degenerative tissue using the Hydrocision TenJet system; Device: Hydrocision Tenjet System
- Shoulder Calcific Tendinosis (Calcific Shoulder Tendinopathy): Treatment of participants diagnosed with Calcific Shoulder Tendinopathy
  Interventions: Procedure: Resection (removal) of the degenerative tissue using the Hydrocision TenJet system; Device: Hydrocision Tenjet System

INTERVENTIONS:
Procedure: Resection (removal) of the degenerative tissue using the Hydrocision TenJet system — During the procedure, the TenJet device will remove degenerative tendinopathic tissue using pressurized saline without causing harm to the healthy tendon fibers.
Device: Hydrocision Tenjet System — The TenJet system will be used during surgery to remove the damaged tissue from the joint

SUMMARY:
Treatment of recalcitrant tendinopathy remains a clinical challenge for physicians without a minimally invasive treatment option that can consistently provide patients with a long-term relief from chronic pain and ability to return to function.

Surgical debridement of degenerative tendon tissue has long been the standard of care to treat degenerative tendon pathology once all conservative or minimally invasive treatment options have failed.

Ultrasound guided tenotomy is an emerging treatment option with the potential to address the underlying degenerative, diseased tissue, by selectively resecting and removing the tissue in a minimally invasive manner. Additionally, with the availability of in-office diagnostic ultrasound imaging, physicians now have an opportunity to evaluate and classify underlying tendon pathology during a clinical exam. This study is to evaluate outcomes in patients presenting with a clinical history of recalcitrant tendinopathy with confirmed diagnosis of degenerative tendinosis using diagnostic ultrasound imaging or MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 - 70 years of age
* Chronic tendon pain ≥ 3 months duration
* History and clinical examination consistent with tendinosis
* Sonographic or MRI confirmation of tendinosis
* 3 months of conservative treatment
* Patient is willing and able to provide informed consent and comply with the study protocol

Exclusion Criteria:

* Full thickness tear of the tendon
* Unable to withhold anticoagulants 7 days prior to the procedure.
* Use above 81mg/day of acetylsalicyclic acid (ASA) and/or non-steroidal anti-inflammatory drug (NSAID) within 7 days of treatment
* Steroid, PRP, Stem cell or biologic injections within 3 months of the study procedure date
* Needle tenotomy, Tenex, or surgical interventions within 6 months of study procedure date
* Active local or systemic infection requiring antiviral, antibacterial or antifungal treatment
* Chronic conditions such as CRPS or fibromyalgia that might affect pain symptoms.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between 18-70 years old presenting with chronic, refractory lateral and medial elbow, hip, or shoulder pain, secondary to tendinosis.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | 2 years
  Using the Visual Analog Scale for Pain (VAS) participants will be asked to report their pain score after surgery
Return to function (Elbow #1) | 2 years
  This will be measured in participants undergoing treatment for Elbow Tendinopathy using the Mayo Elbow Performance Score (MEPS)
Return to function (Elbow #2) | 2 years
  This will be measured in participants undergoing treatment for Elbow Tendinopathy using the Patient-Rated Tennis Elbow Evaluation (PRTEE) survey
Return to function (Elbow #3) | 2 years
  This will be measured in participants undergoing treatment for Elbow Tendinopathy using the Quick Disability Arm, Shoulder and Hand (QDASH) survey
Return to function (All cohorts) | 2 years
  This will be measured in participants undergoing treatment for Elbow, Hip and Shoulder Tendinopathy using the Short Form Health Survey (SF-12) survey
Return to Function (Hip) | 2 years
  This will be measured in participants undergoing treatment for Hip Tendinopathy using the Victorian Institute of Sport Assessment-Gluteal Questionnaire (VISA-G) survey
Return to Function (Shoulder) | 2 years
  This will be measured in participants undergoing treatment for Shoulder Tendinopathy using the American Shoulder & Elbow Score (ASES) survey

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Standford Medicine, Redwood City, California
  - Cleveland Clinic, Coral Springs, Florida
  - Ochsner Health, Baton Rouge, Louisiana
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Lorain, Ohio
  - Penn Highlands Orthopedics and Sports Medicine, Clarion, Pennsylvania
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania